CLINICAL TRIAL: NCT04283045
Title: Community-based Adaptive Autism Intervention for Toddlers
Acronym: CAIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Connie Kasari, Ph.D., Professor/PhD, University of California, Los Angeles
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-000197
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD; autism; JASPER; JASPER Plus+
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Activator Appliances

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JASPER (6 weeks) (Active Comparator): Child will be randomized to spend an hour daily, 5 days a week with teaching assistant (TA) doing JASPER for the following 6 weeks. If child is an early responder, he/she will continue to do JASPER daily, 5 times a week, for the remaining 18 weeks of the study.
  If child is a slow responder, he/she can get randomized to receive 30 minutes of JASPER Plus+ and 30 minutes of JASPER with a TA daily, 5 days a week for the remaining 18 weeks of the study.
  Or
  Child can get randomized to continue his/her daily sessions of JASPER with the TA for an hour each day, 5 days a week for the following 18 weeks of the study.
  Interventions: Behavioral: JASPER; Behavioral: JASPER Plus+
- JASPER (12 weeks) (Active Comparator): Child will be randomized to spend an hour daily, 5 days a week with teaching assistant (TA) doing JASPER for the following 12 weeks. If child is an early responder, he/she will do JASPER for 60 minutes with TA, 5 times a week, for the remaining 12 weeks of the study.
  If child is a slow responder, he/she can get randomized to receive 30 minutes of JASPER Plus+ and 30 minutes of JASPER with a TA daily, 5 days a week for the remaining 12 weeks of the study.
  Or
  Child can get randomized to continue his/her daily sessions of JASPER with the TA for an hour each day, 5 days a week for the following 12 weeks of the study.
  Interventions: Behavioral: JASPER; Behavioral: JASPER Plus+

INTERVENTIONS:
Behavioral: JASPER — JASPER is a developmentally anchored behavioral intervention that assumes that communication develops from social interactions in which specific social engagement strategies, symbolic representations, and early communication forms are modeled and naturally reinforced by the adult's responses to the child. The adult referred in this condition is the TA.
Behavioral: JASPER Plus+ — JASPER Plus+ refers to direct instruction of social communication targets of pointing to share, showing gesures, and give to share gestures, and play targets at the child's target play level.
  JASPER Plus+ will occur at a table top with repeated trials of instruction until the child can produce the desired behavior on their own.

SUMMARY:
The proposed study (CAIT: Community-based Adaptive Autism Intervention for Toddlers) aims to determine the most optimal sequence of interventions for improving the social- communicative, language and cognitive outcomes of toddlers with autism spectrum disorder (ASD). The target population consists of 2-3 year-old children with ASD who receive community based, publicly funded early intervention in two authentic educational settings in East Harlem and the Bronx, NY known as New York Center for Infants & Toddlers (NYCIT). An expected 300 toddlers with ASD will participate with their community-recruited paraprofessional teaching assistants (TAs) and group leaders (GLs). The study aims to construct the most effective one-year, two-phase, adaptive intervention, in which intervention is individualized based on a child's initial response to intervention. Phase 1, from program entry to either 6 or 12 weeks (randomized), involves 60 minutes daily of an evidence based social communication intervention, JASPER (Joint Attention, Symbolic Play, Engagement & Regulation) delivered 1-on-1 to the child by the trained TA. At end of Phase 1, response to intervention is rated by the GLs for slow or fast improvements of joint engagement (a core deficit in the early development of children with ASD, and a significant indicator of good progress toward improving social communication and language). In Phase 2 (to week 24), toddlers responding slowly are re-randomized to continue with JASPER for 60 minutes per day or augment treatment with direct, structured teaching of social communication targets for 30 minutes and JASPER for another 30 minutes per day. Toddlers responding quickly are given 30 minutes of JASPER and 30 minutes of jasPEER (JASPER with a peer) to further improve socialization and social communication.

DETAILED DESCRIPTION:
This study will use a Sequential Multiple Assignment Randomized Trial (SMART) design to assess when to examine initial response to treatment, as well as whether and how best to augment the current first line, standard of care intervention for children demonstrating a slower response.

First, at program entry, the investigators will assess all toddlers using both standardized and experimental assessments as they enroll in the NYCIT program. After entry assessments, the investigators will randomize each child with equal probability to early response assessment at either six weeks or 12 weeks (timing). This early response assessment will be used to determine whether children are considered fast or slow responders to treatment. Children who are considered early responders will continue to receive JASPER. Children responding slowly to the initial intervention will be randomized to continue JASPER or to add JASPER Plus+ to their JASPER sessions. Approximately 200-300 toddlers (24-36 months) with a diagnosis of ASD, as confirmed by clinical evaluation records required for placement at the NYCIT will participate. Children will be assessed prior to intervention, immediately after Stage 1(early response) at either six or twelve weeks, exit Stage 2 intervention, and follow up.

If teacher/paraprofessional withdraws from the study, all reasonable efforts will be made to place the child with another consenting teacher/paraprofessional. Based on the first two years of trials working with this center, no teacher withdrew mid study. However, a small number of teachers did change positions or took leave (e.g., maternity leave, move for job in another district). In these cases, the child was transferred to another consenting teacher.

SMART Design:

Initial Randomize to Stage 1 Treatment

Stage 1: JASPER (6 weeks)

Early Responders/Slow Responders determined

Stage 2: JASPER (Early Responders only)-A

Slow Responders randomized to Stage 2: JASPER Plus+ + JASPER -B or Stage 2: JASPER (Randomized for slow responders)-C A, B, and C options occur during the following 18 weeks

Exit assessments and Follow up assessments at 3 months post exit

Initial Randomized to Stage 1 Treatment

Stage 1: JASPER (12 weeks)

Early Responders/Slow Responders determined

Stage 2: JASPER (Early Responders only)- D Slow Responders randomized to Stage 2: JASPER Plus+ + JASPER - E or Stage 2: JASPER (Randomized for slow responders)- F D, E, and F options occur during the following 12 weeks

ELIGIBILITY:
Child Inclusion Criteria:

* diagnosis of ASD based on clinical report or ADOS-2 if needed
* chronological age less than 36 months
* caregiver consent to learn intervention strategies if randomized to either parent condition.

Exclusion Criteria:

* Child has co-morbid disorders such as cerebral palsy or down syndrome.

Ages: 24 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 199 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in social communicative utterances (SCU) using Short Play and Communication Evaluation (SPACE) | entry (1st month of study) and 6 weeks after entry
  The assessment is delivered in the context of play and takes approximately 15 minutes. The change in number of socially communicative utterances (SCU) will be recorded as primary outcome.
Change in social communicative utterances (SCU) using Short Play and Communication Evaluation (SPACE) | 6 weeks after entry and 12 weeks after entry
  The assessment is delivered in the context of play and takes approximately 15 minutes. The change in number of socially communicative utterances (SCU) will be recorded as primary outcome.
Change in social communicative utterances (SCU) using Short Play and Communication Evaluation (SPACE) | 12 weeks after entry and 24 weeks after entry
  The assessment is delivered in the context of play and takes approximately 15 minutes. The change in number of socially communicative utterances (SCU) will be recorded as primary outcome.
Change in social communicative utterances (SCU) using Short Play and Communication Evaluation (SPACE) | 24 weeks after entry and 3 months after intervention (36 weeks)
  The assessment is delivered in the context of play and takes approximately 15 minutes. The change in number of socially communicative utterances (SCU) will be recorded as primary outcome.
Change in social communicative utterances (SCU) using JASPER Deployment Project Treatment Fidelity Checklist (TCX) | entry (1st month of study) and 6 weeks after entry
  The assessment is delivered in the context of play and takes approximately 15 minutes. The change in number of socially communicative utterances (SCU) will be counted as the primary outcome.
Change in social communicative utterances (SCU) using JASPER Deployment Project Treatment Fidelity Checklist (TCX) | 6 weeks after entry and 12 weeks after entry
  The assessment is delivered in the context of play and takes approximately 15 minutes. The change in number of socially communicative utterances (SCU) will be counted as the primary outcome.
Change in social communicative utterances (SCU) using JASPER Deployment Project Treatment Fidelity Checklist (TCX) | 12 weeks after entry and 24 weeks after entry
  The assessment is delivered in the context of play and takes approximately 15 minutes. The change in number of socially communicative utterances (SCU) will be counted as the primary outcome.
Change in social communicative utterances (SCU) using JASPER Deployment Project Treatment Fidelity Checklist (TCX) | 24 weeks after entry and 3 months after intervention (36 weeks)
  The assessment is delivered in the context of play and takes approximately 15 minutes. The change in number of socially communicative utterances (SCU) will be counted as the primary outcome.

SECONDARY OUTCOMES:
Change in play levels/types using the Short Play and Communication Evaluation (SPACE) | entry (1st month of study) and 6 weeks after entry
  The change in different play types and play level will be used as secondary outcome throughout the study.
Change in play levels/types using the Short Play and Communication Evaluation (SPACE) | 6 weeks after entry and 12 weeks after entry
  The change in different play types and play level will be used as secondary outcome throughout the study.
Change in play levels/types using the Short Play and Communication Evaluation (SPACE) | 12 weeks after entry and 24 weeks after entry
  The change in different play types and play level will be used as secondary outcome throughout the study.
Change in play levels/types using the Short Play and Communication Evaluation (SPACE) | 24 weeks after entry and 3 months after intervention (36 weeks)
  The change in different play types and play level will be used as secondary outcome throughout the study.
Change in joint engagement using the JASPER Deployment Project Treatment Fidelity Checklist (TCX) | entry (1st month of study) and 6 weeks after entry
  The assessment is delivered in the context of play and takes approximately 15 minutes. The change in joint engagement will be used as secondary outcome.
Change in joint engagement using the JASPER Deployment Project Treatment Fidelity Checklist (TCX) | 6 weeks after entry and 12 weeks after entry
  The assessment is delivered in the context of play and takes approximately 15 minutes. The change in joint engagement will be used as secondary outcome.
Change in joint engagement using the JASPER Deployment Project Treatment Fidelity Checklist (TCX) | 12 weeks after entry and 24 weeks after entry
  The assessment is delivered in the context of play and takes approximately 15 minutes. The change in joint engagement will be used as secondary outcome.
Change in joint engagement using the JASPER Deployment Project Treatment Fidelity Checklist (TCX) | 24 weeks after entry and 3 months after intervention (36 weeks)
  The assessment is delivered in the context of play and takes approximately 15 minutes. The change in joint engagement will be used as secondary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- New York Center for Infants and Toddlers, Inc., New York, New York, United States

REFERENCES:
- [Derived] Shire SY, Shih W, Chang YC, Kodjoe M, Nodzo S, Kasari C. Comparing the Implementation Context for Early Intervention Services Before and During the COVID-19 Pandemic. Prev Sci. 2024 Jun 11. doi: 10.1007/s11121-024-01696-5. Online ahead of print. PMID 38862831